CLINICAL TRIAL: NCT04633616
Title: Tailored Patient-Provider Communication (TPPC): A Pragmatic Single-Blinded Trial Evaluating the Impact of TPPC in Dermatology Patients Compared to Standard Patient-Provider Communication.
Brief Title: Tailored Patient-Provider Communication (TPPC): Evaluating the Impact of TPPC in Dermatology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Psoriasis Foundation (Other)
Responsible Party: Principal Investigator, April Armstrong, Doctor/Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: APP-18-03588
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Psoriasis; Atopic Dermatitis; Acne
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Tailored patient-provider communication versus non-tailored patient-provider communication on patient recruitment to clinical trials and patient engagement.
Who Masked: Care Provider, Investigator
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored Delivery of Education (Experimental): Communication will be tailored as the mode of weblink delivery will be customized to patient preference.
  Interventions: Other: Tailored Patient-Provider Communication
- Non-tailored Delivery of Education (Placebo Comparator): Communication will be non-tailored such that patients will not be able to choose their preferred mode of communication and will receive hardcopy.
  Interventions: Other: Non-Tailored Patient-Provider Communication

INTERVENTIONS:
Other: Tailored Patient-Provider Communication — Every 1.5 months, patients randomized to the tailored patient-provider communication model will receive weblinks directing patients to disease-specific educational videos and associated questionnaires. Communication will be tailored as the mode of weblink delivery will be customized to patient preference. Patients can choose messages to be delivered via e-mail, SMS, WhatsApp, or Facebook. For example, if one patient determines SMS messaging as their preferred communication mode, then this patient will receive a weblink via SMS directing the patient to customized educational videos and questionnaires. Weblinks delivered via tailored patient-provider communication will be enabled by Wecudos.
  Arms: Tailored Delivery of Education
Other: Non-Tailored Patient-Provider Communication — Every 1.5 months, patients randomized to the non-tailored patient-provider communication model will receive weblinks directing patients to disease-specific educational videos and associated questionnaires. Communication will be non-tailored such that patients will not be able to choose their preferred mode of communication and will receive hardcopy. Patients will receive hardcopy on how to access psoriasis education. Weblinks delivered via non-tailored patient-provider communication will be enabled by Wecudos.
  Arms: Non-tailored Delivery of Education

SUMMARY:
The impact of tailored patient-provider communication to improve clinical trial recruitment, patient knowledge, and patient engagement will be studied. Tailored patient-provider communication refers to the individualization of patient-provider communication using patients' preferred methods of communication. This involves the utilization of social messaging such as e-mail or text and/or social media platforms. These communication methods purport to and meet individual patient needs whilst ensuring that information is received and in a format that is familiar to each patient. The primary outcomes of the proposed research is to evaluate the impact of tailored patient-provider communication on patient response rates (speed and number), clinical trial recruitment rates, patient knowledge, and patient engagement.

DETAILED DESCRIPTION:
This is a 3-month, pragmatic, single-blinded randomized controlled trial evaluating the impact of tailored patient-provider communication on patient engagement and clinical outcomes of adult dermatology patients compared to non-tailored patient-provider communication. The pragmatic trial will compare patient engagement and clinical outcomes between the two models. The rationale for proposing a pragmatic trial is to test whether tailored patient-provider communication works in real life. This design allows for a large spectrum of everyday clinical settings in order to maximize applicability and generalizability. The pragmatic approaches are especially pronounced along the inclusive eligibility criteria, experimental intervention flexibility, and primary outcome being highly relevant to patients and providers alike.

The investigators will recruit from approximately 32,310 adult patients from target populations, southern California to enroll 134 participants in the study. In addition to recruiting from the general population, the investigators will place a specific emphasis on recruiting patients living in rural and underserved communities; the investigators will also recruit from a full range of dermatological diseases.

Patient recruitment and enrollment will begin the first month of year one and continue through the fourth month of year one. The expected duration of this pragmatic, single-blinded randomized controlled equivalency trial for each participant will be a maximum of 3 months, including an initial baseline visit. No additional follow-up visits beyond this are expected for this research study.

Patients will be randomized to receive patient education via tailored or non-tailored patient-provider communication. The study team will know which form of communication each patient will receive while study participants will not know the different types of communication being studied. Patients randomized to either study population groups can be assessed remotely or in-person at the screening/baseline visit. At month 3, all patients will take high-quality photographs of their skin and submit these pictures to our dermatologist online. Any additional in-person or remote visits will be determined by providers and patients just as they would occur in the real-world. Primary and secondary outcomes will be monitored at months 0, 1.5, and 3.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Speak English or Spanish
* Male or female, at least 18 years of age
* Have an active, physician-diagnosed dermatological condition
* Have access to an electronic device that is capable of capturing images with a minimum resolution of 1024x768 pixels
* Have access to at least one form of social messaging (e-mail, SMS, WhatsApp, or Facebook) which can connect online

Exclusion Criteria:

* Does not have an active dermatological condition at the beginning of the study
* Does not live in southern California
* Unable to fulfill the required tasks of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Patient Response Rates | 3 months
  Patient response rate will determine the first step of patient engagement and assesses a patients willingness to 'interact' with the weblink delivered. Patient response rates will be measured by click rates. Click rates will be calculated using the proportions of patients in both study populations who choose to click on the weblinks delivered throughout the study, regardless of whether or not questionnaires are completed. The time elapsed from when the weblink is sent and when the weblink is clicked will also be recorded.

SECONDARY OUTCOMES:
Patient Activation | 3 months
  Measured by the proportion of patients achieving patient activation level 3 or 4 on the Patient Activation Measure 13-item measurement (PAM-13). The PAM-13 score is a validated scale consisting of 13 questions that will determine patient 'activation', or 'empowerment' of a patient to participate in their healthcare. The higher the score, the higher the activation level. Patients in level 1 may still believe their nurse or doctor will "fix" them. Patients in level 2 may understand they must be involved in their healthcare but lack the knowledge and confidence to take care of their conditions. Patients in level 3 are beginning to gain confidence to take on self-management behaviors and need to experience small successes to build a sense of self-efficacy and increase activation. Patients in level 4 have the confidence and skills to manage their health but may need help with maintaining their progress during stressful times.
Patient Experience | 3 months
  Measured by the proportion of patients who report 'good' or 'very good' on the Armstrong Viewer Assessment (AVA). The AVA is a validated scale that will be used to determine patient experience with the educational materials viewed. Patients will be asked to complete this single question questionnaire after watching each educational video. This will ask how each participant felt about the video using a 5-point Likert scales between 0-4, where 0=very poor, 1=poor, 2=fair, 3=good, and 4=very good.
Patient Drop-out Rate | 3 months
  Patient drop-out rate will determine the proportion of patients who 'accept' the delivered weblinks.

OTHER OUTCOMES:
Potential clinical trial recruitment rate | 3 months
  Potential clinical trial recruitment rate will be descriptively assessed in patients who are sent educational content pertaining to clinical trial opportunities via weblinks.
Patient Knowledge | 3 months
  Patient knowledge after watching educational materials will be measured in two ways: 1) patients' perceived knowledge, and 2) patients' actual knowledge. First, patients' perceived knowledge will be assessed using a single question questionnaire. The weblink delivered to patients will direct patients to this questionnaire. This will ask what each participant perceived their knowledge levels to be regarding the video content using a 5-point Likert scale between 0-4, where 0=very poor, 1=poor, 2=fair, 3=good, and 4=very good. This questionnaire typically takes 10-20 seconds to complete. Second, patients' actual knowledge will be assessed using customized 5-question questionnaires. The weblink delivered to patients will direct patients to this questionnaire. This will ask each participant 5 customized questions relating to the educational material viewed.

CONTACTS AND LOCATIONS:
Overall Officials: April Armstrong, MD, MPH, Principal Investigator — University of Southern California
Locations (1):
- USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Subject confidentiality is strictly held in trust by the investigators, study staff, and the sponsor(s) and their agents. The study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.
  The study monitor or other authorized representatives of the sponsor may inspect all study documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) for the study subjects. The clinical study site will permit access to such records.